CLINICAL TRIAL: NCT06285318
Title: A Retrospective, Multicountry Study of Clinical Outcomes in Patients With Relapsed/Refractory Multiple Myeloma Treated With T-cell Redirectors Outside of Clinical Trials
Brief Title: A Study of Clinical Outcomes in Patients With Relapsed/Refractory Multiple Myeloma (RRMM) Treated With T-cell Redirectors Outside of Clinical Trials
Acronym: REALiTEC/TAL
Status: Recruiting | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 64007957MMY4004; 64007957MMY4004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2023-11-27; First posted 2024-02-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Multiple Myeloma (RRMM)
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Participants with Relapsed/Refractory Multiple Myeloma (RRMM): Teclistamab Cohort 1: Participants with RRMM who received at least one dose of teclistamab outside of clinical trials on or before 31 December 2022 will be enrolled in the study. The data available from the medical records of each enrolled participant will be the collected to describe the use of teclistamab.
  Interventions: Other: Teclistamab
- Participants with Relapsed/Refractory Multiple Myeloma (RRMM): Teclistamab Cohort 2: Participants with RRMM who received at least one dose of teclistamab outside of clinical trials from 01 January 2023 to 31 December 2024, inclusive will be enrolled in the study. The data available from the medical records of each enrolled participant will be the collected to describe the use of teclistamab.
  Interventions: Other: Teclistamab
- Participants with RRMM: Teclistamab Cohort 3: Participants with RRMM who received at least one dose of teclistamab outside of clinical trials from 01 January 2025 to 31 December 2025, inclusive will be enrolled in the study. The data available from the medical records of each enrolled participant will be the collected to describe the use of teclistamab.
  Interventions: Other: Teclistamab
- Participants with RRMM: Talquetamab Cohort: Participants with RRMM who received at least one dose of talquetamab outside of clinical trials on or before 31 December 2023 will be enrolled in the study. The data available from the medical records of each enrolled participant will be collected to describe the use of talquetamab.
  Interventions: Other: Talquetamab

INTERVENTIONS:
Other: Teclistamab — No Intervention will be administered during the study. Retrospective data analysis using participants medical records collected within this study will be entered into CRF.
  Other Names: TECVAYLI
  Groups: Participants with RRMM: Teclistamab Cohort 3; Participants with Relapsed/Refractory Multiple Myeloma (RRMM): Teclistamab Cohort 1; Participants with Relapsed/Refractory Multiple Myeloma (RRMM): Teclistamab Cohort 2
Other: Talquetamab — No Intervention will be administered during the study. Retrospective data analysis using participants medical records collected within this study will be entered into CRF.
  Other Names: TALVEY
  Groups: Participants with RRMM: Talquetamab Cohort

SUMMARY:
The purpose of this study is to describe the use of teclistamab/talquetamab in the treatment of patients with RRMM outside of clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented diagnosis of multiple myeloma
* Received the first dose of teclistamab on or before 31 December 2022, regardless of the duration of teclistamab treatment (REALiTEC cohort 1) OR Received the first dose of teclistamab from 01 January 2023 to 31 December 2024, inclusive, regardless of the duration of teclistamab treatment (REALiTEC cohort 2) OR Received the first dose of teclistamab from 01 January 2025 to 31 December 2025, inclusive, regardless of the duration of teclistamab treatment (REALiTEC cohort 3) OR Received the first dose of talquetamab on or before 31 December 2023, regardless of the duration of talquetamab treatment (REALiTAL cohort). Participants who received both teclistamab & talquetamab can be included in both REALiTEC and REALiTAL cohorts
* Received at least one dose of teclistamab/talquetamab
* Provision of a patient-signed informed consent form (ICF), or an ICF waiver for deceased patients as applicable based on country/site-specific requirements

Exclusion Criteria:

* To be excluded from REALiTEC cohorts if received teclistamab as part of an interventional clinical trial
* To be excluded from REALiTAL cohort if received talquetamab as part of an interventional clinical trial
* Participants who have received teclistamab as part of a Janssen pre-approval access program are excluded from the REALiTEC Cohort 2 and REALiTEC Cohort 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population include patients who have initiated the treatment with T-cell redirectors outside of a clinical trial setting.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Describe Baseline Characteristics of Participants with Relapsed/Refractory Multiple Myeloma (RRMM) who Received Teclistamab/ Talquetamab Outside of Clinical Trials | Baseline (Day 1)
  Participants' demographics and disease characteristics (age, co-morbidities, renal function), and prior antimyeloma therapies will be reported.
Overall Response Rate (ORR) in Participants with RRMM who Received Teclistamab/Talquetamab Outside of Clinical Trials | Up to 40 months
  ORR is defined as the percentage of patients who have a PR or better as assessed by investigator per International Myeloma Working Group (IMWG) response criteria.
Time to First Response in Participants with RRMM who Received Teclistamab/Talquetamab Outside of Clinical Trials | Up to 40 months
  Time to first response is defined as the time between date of first dose of teclistamab/talquetamab and the date when patient has achieved first response, as assessed by investigator per IMWG response criteria.
Time to Best Response in Participants with RRMM who Received Teclistamab/Talquetamab Outside of Clinical Trials | Up to 40 months
  Time to best response is defined as the time between date of first dose of teclistamab/talquetamab and the date of the best response, as assessed by investigator per IMWG response criteria.
Duration of Response (DOR) in Participants with RRMM who Received Teclistamab/Talquetamab Outside of Clinical Trials | Up to 40 months
  DOR will be calculated among participants (with a PR or better response) from the date of the first response (PR or better) to the date of first evidence of progressive disease, as assessed by investigator per IMWG response criteria.
Minimal Residue Assessment (MRD) in Participants with RRMM who Received Teclistamab/Talquetamab Outside of Clinical Trials | Up to 40 months
  Number of participants with MRD negative rate will be assessed.
Overall Survival (OS) in Participants with RRMM who Received Teclistamab/Talquetamab Outside of Clinical Trials | From the date of first dose of teclistamab/talquetamab to the date of the participant's death (up to 40 months)
  OS is defined as the time from the date of first dose of teclistamab/talquetamab to the date of the participant's death.
Progression Free Survival (PFS) in Participants with RRMM who Received Teclistamab/Talquetamab Outside of Clinical Trials | Up to 40 months
  PFS is defined as the time from the date of first dose of teclistamab/talquetamab to the date of first evidence of progressive disease, as assessed by investigator per IMWG response criteria, or death due to any cause, whichever occurs first.
Time to Next Treatment (TTNT) in Participants with RRMM who Received Teclistamab/Talquetamab Outside of Clinical Trials | Up to 40 months
  TTNT is defined as the time from the date of first dose of teclistamab/talquetamab to the start of the next line of antimyeloma treatment.
Describe the Safety Management of Teclistamab/Talquetamab in the Treatment of Participants with RRMM Outside of Clinical Trials | Baseline (Day 1) up to end of treatment (up to 40 months)
  Incidence and severity of adverse events (AEs) including immune effector cell-associated neurotoxicity syndrome (ICANS), cytokine release syndrome (CRS) and other AEs as well as medications used for prophylaxis and management of adverse events will be reported.

SECONDARY OUTCOMES:
Describe the Use of Teclistamab/Talquetamab in the Treatment of Participants with RRMM Outside of Clinical Trials | Baseline (Day 1) up to end of treatment (up to 40 months)
  Treatment patterns including healthcare setting and treatment schedules will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Limited Clinical Trial, Study Director — Janssen-Cilag Limited
Locations (68):
- Denmark (5):
  - Aalborg Sygehus Syd, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
  - Sygehus Lillebælt, Vejle, Vejle
- France (6):
  - Hopital Albert Calmette - CHU Lille, Lille
  - Institut Paoli Calmettes, Marseille
  - CHU de Nantes hotel Dieu, Nantes
  - Hopital Saint Louis, Paris
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - CHRU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (7):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - University Hospital Hamburg Eppendorf, Hamburg
  - Klinikum Region Hannover Klinikum Siloah, Hanover
  - Uniklinikum Heidelberg, Heidelberg
  - Klinikum Nurnberg Nord, Nuremberg
  - Universitätsklinikum Würzburg Med. Klinik U. Poliklinik Ii, Würzburg
- Greece (9):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Laiko General Hospital of Athens, Athens
  - Alexandra Hospital, Athens
  - University Hospital of Crete, PAGNI, Heraklion
  - Ioannina University Hospital, Ioannina
  - University Hospital Of Larissa, Larissa
  - Anticancer Hospital of Thessaloniki Theageneio, Thessaloniki
  - Ahepa University General Hospital of Thessaloniki, Thessaloniki
  - G Papanikolaou Hospital of Thessaloniki, Thessaloniki
- Ireland (5):
  - Cork University Hospital, Cork
  - Bon Secours Hospital, Cork
  - St James Hospital, Dublin
  - Beacon Hospital, Dublin
  - University Hospital Galway - Ireland, Galway
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (16):
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Sanitaria dell'Alto Adige - Ospedale di Bolzano, Bolzano
  - Ospedale A.Perrino di Brindisi, Brindisi
  - AOU Careggi, Florence
  - Ospedale Vito Fazzi, Lecce
  - Policlinico di Milano, Milan
  - IRCCS Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Casa di Cura La Maddalena, Palermo
  - Universita Cattolica del Sacro Cuore - Fondazione Policlinico Universitario 'A. Gemelli', Roma
  - Presidio Ospedaliero Santo Spirito in Sassia, Roma
  - Ospedale Andrea Tortora Pagani Salerno, Salerno
  - Ospedale Ca' Foncello, Treviso
  - Azienda Sanitaria Universitaria Giuliano Isontina Ospedale Maggiore, Trieste
  - Ospedale Castelli, Verbania
  - Ospedale San Bortolo, Vicenza
- Norway (2):
  - Akershus Universitetssykehus, Oslo
  - Vestfold Hospital Trust, Tønsberg
- Spain (7):
  - Hosp. Ntra. Sra. de Sonsoles, Ávila
  - Hosp. Univ. Virgen de Las Nieves, Granada
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. de La Paz, Madrid
  - Hosp. Costa Del Sol, Málaga
  - Hosp. Clinico Univ. de Valencia, Valencia
  - Hosp. Alvaro Cunqueiro, Vigo
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Länssjukhuset Ryhov, Jönköping
  - Karolinska Universitetssjukhuset, Stockholms
  - Uddevalla Hospital, Uddevalla
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - University College Hospital, London
  - Guys and St Thomas NHS Foundation Trust, London
  - The Royal Wolverhampton Hospitals NHS Trust - New Cross Hosp, Wolverhampton

IPD SHARING:
Plan to Share IPD: No